CLINICAL TRIAL: NCT01620307
Title: Adjuvant Treatment With a mTOR Inhibitor, Rapamune Improves Outcomes of Severe H1N1 Pneumonia With Acute Respiratory Failure
Brief Title: Rapamune Improves Outcomes of Severe H1N1 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung Fu-Tsai, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB:100-2433C
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: H1N1 Pneumonia; Hypoxemia
Keywords: H1N1 patients with severe hypoxemia requiring ventilator support
MeSH Terms: conditions — Hypoxia | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with Rapamune treatment (Active Comparator): All patients were treated with Oseltamivir (Tamiflu, Roche) 50 mg twice a day for 10 days and oral prednisolone 20 mg/day for 14 days. At ICU admission, patients started on empiric antimicrobial therapy with moxifloxacin 500 mg per day until results of microbiological studies were available.
  Each patient received best support treatment including mechanical ventilator, fluid resuscitation, gastrointestinal and thromboembolic prophylaxis, and enteral nutrition for most aspects of care. After radomization, patients were received Sirolimus (Rapamune 2mg/day, Pfizer)for a course of 14 days.
  Interventions: Drug: Sirolimus (Rapamune 2mg/day, Pfizer)
- Without Rapamune treatment. (Placebo Comparator): All patients were treated with Oseltamivir (Tamiflu, Roche) 50 mg twice a day for 10 days and oral prednisolone 20 mg/day for 14 days. At ICU admission, patients started on empiric antimicrobial therapy with moxifloxacin 500 mg per day until results of microbiological studies were available.
  Each patient received best support treatment including mechanical ventilator, fluid resuscitation, gastrointestinal and thromboembolic prophylaxis, and enteral nutrition for most aspects of care. After radomization, patients were not to receive Sirolimus (Rapamune 2mg/day, Pfizer)for a course of 14 days.
  Interventions: Drug: Sirolimus (Rapamune 2mg/day, Pfizer)

INTERVENTIONS:
Drug: Sirolimus (Rapamune 2mg/day, Pfizer) — Sirolimus (Rapamune 2mg/day, Pfizer) or not for a course of 14 days.

SUMMARY:
Severe H1N1 pneumonia with acute respiratory failure shows hyperactive immune cells infiltration of lung. Rapamune, a mTOR inhibitor, modulates the immune response by blocking activation of T- and B-cells. To investigate the clinical efficiency of rapamune in severe H1N1 pneumonia with respiratory failure, this study was conducted.

DETAILED DESCRIPTION:
From 2009 winter to 2011 spring, patients with flu-like symptoms in Chang Gung Memorial Hospital were screened by rapid antigen test and influenza subtype was confirmed by polymerization chain reaction (PCR). 38 H1N1 patients with severe hypoxemia [alveolar-arterial oxygen gradient, (A-a) O2 gradient, > 200 mmHg] requiring ventilator support were randomized to receive Rapamune (2mg/day) or not. Patients were then randomized to receive either Sirolimus (Rapamune 2mg/day, Pfizer) or not for a course of 14 days. The outcome variables include liberation of ventilator, ICU mortality, necessity of ECMO, Sequential Organ Failure Assessment (SOFA) score and complications after admission to ICU were recorded. SOFA score composed of scores from six organ systems, graded from 0 to 4 according to the degree of dysfunction/failure.

ELIGIBILITY:
Inclusion Criteria:

* H1N1 patients with severe hypoxemia [alveolar-arterial oxygen gradient, (A-a) O2 gradient, > 200 mmHg] requiring ventilator support were included to randomization.

Exclusion Criteria:

* severity of illness and multiple organ dysfunction (MOD) were assessed within 24 hours of ICU admission.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
liberation of ventilator | 28 days
  Patients were then randomized to receive either Sirolimus (Rapamune 2mg/day, Pfizer) or not for a course of 14 days. Ventilator management was previously described. The ventilator liberation rate is primary outcome.

SECONDARY OUTCOMES:
necessity of Extracorporeal membrane oxygenation(ECMO) | 28 days
  Patients were then randomized to receive either Sirolimus (Rapamune 2mg/day, Pfizer) or not for a course of 14 days. Ventilator management was previously described.Extracorporeal membrane oxygenation (ECMO) was used in patients with severe refractory hypoxemia

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Chang Gung Memorial Hospital